CLINICAL TRIAL: NCT01288053
Title: Non-myeloablative Allogeneic Hematopoietic Stem Cell Transplantation (NST) for Patients With Refractory Crohn's Disease
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: No participant enrolled more than two years. No plan to continue study.
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Richard Burt, MD, MD, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DIADCDAllo2005
Record Dates: First submitted 2011-01-27; First posted 2011-02-02 (Estimated); Results first posted 2018-08-06 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Allogeneic Stem Cell Therapy (Experimental): Allogeneic Stem Cell Therapy will be performed after conditioning
  Interventions: Biological: Allogeneic Stem Cell Therapy

INTERVENTIONS:
Biological: Allogeneic Stem Cell Therapy — Donor stem cells will be given to subject diagnosed with Crohn's disease

SUMMARY:
Allogeneic transplantation has been a high-risk procedure, although non-myeloablative conditioning regimens (mini-transplantation) minimizes regimen related toxicity. The investigators, therefore, propose a phase I study of matched sibling allogeneic hematopoietic stem cell transplantation with non-myeloablative conditioning. In addition, graft versus host disease (GVHD) will be virtually eliminated by CAMPATH that removes donor T cells from the graft.

The goal is to assess the toxicity/efficacy (phase I) of allogeneic non-myeloablative hematopoietic stem cell transplantation for high-risk Crohn's disease. In simplistic terms, this protocol is designed to ablate an aberrant immune system and then, similar to the use of marrow transplants for immunodeficient patients, reconstitute a new immune system with lymphocyte depleted marrow.

DETAILED DESCRIPTION:
PBSC will be mobilized with G-CSF 10 mcg/kg/day (dose may be adjusted down to 5 mcg/kg/day by PI for toxicity, e.g. flu-like symptoms) with stem cell collection beginning on day 4 or 5. Leukapheresis may be repeated up to three consecutive days.

Cyclophosphamide 60 mg/kg/day x 2 days will be given IV over 1 hour in 500 cc of normal saline.

Dosage should be based on the lesser of adjusted body weight or actual weight. Mesna 50mg/day x 2 days will be given IV over 24 hours

CAMPATH-1H 30mg/day x 2 days (no dose adjustment) will be given IV over 2 hours in 100 cc of normal saline. Premedication with Solumedrol 1g IV, Acetaminophen 650mg & benadryl 50mg PO/IV will be given 30-60min before infusion. Also while on CAMPATH, Chlorphenamine 4 mg PO TID, Singular 10 mg PO daily, Pepcid 40 mg PO BID and Claritin 10 mg PO daily will be given, adjusted as needed. These medications can be repeated or changed as needed.

Fludarabine 30mg/m2 daily for 3 days (no dose adjustment) will be given IV over 30 minutes in 100 cc normal saline.

Hydration approximately 150ml/hr should begin 2 hours before cyclophosphamide and continue until 24 hours after the last cyclophosphamide dose. Daily weights will be obtained. Amount of fluid can be modified based on patient's fluid status.

G-CSF will be continued until absolute neutrophil count reaches at least 1,000/ul.

Cyclosporin will be started on day -2 at 200 mg po BID and adjusted by HPLC levels to between 150 - 250 or by toxicity (e.g., tremor, renal insufficiency, TTP, etc.). CSA will be continued for 30 days unless stopped for toxicity or needed to maintain donor engraftment.

Cyclosporine and MMF guidelines dosage and duration can be modified according to investigators discretion based on side effects, renal function, CBC and GVHD status.

ELIGIBILITY:
Patient eligibility

Inclusion Criteria:

1. Age >18 years and less than age 45 years at time of pretransplant evaluation and,
2. Ability to give informed consent.

And either A or B A)An established clinical diagnosis of severe CD with disease onset before 16 years old (at least 71 genetic loci predispose to pediatric CD, Limbergen, JV. Annu. Rev. Genom. Human Genet. 2009; 10:89-116) that has failed therapy with prednisone, 5 ASA products and has failed an anti-TNF therapy. Failure is defined as a CDAI (appendix A) 250-400 or a Craig Severity Score that is > 17 (appendix C).

B)Relapse after an autologous HSCT with a CDAI (appendix A) 250-400 or a Craig Severity Score that is > 17 (appendix C).

Exclusion Criteria:

1. HIV positive.
2. History of coronary artery disease, or congestive heart failure.
3. Uncontrolled diabetes mellitus or any other illness that in the opinion of the investigators would jeopardize the ability of the patient to tolerate aggressive chemotherapy.
4. Prior history of malignancy except localized basal cell or squamous skin cancer. Other malignancies for which the patient is judged to be cured by local surgical therapy, such as head and neck cancer, or stage I breast cancer will be considered on an individual basis
5. Positive pregnancy test, lactation, inability or unwillingness to pursue effective means of birth control, failure to accept or comprehend irreversible sterility as a side effect of therapy.
6. Psychiatric illness or mental deficiency making compliance with treatment or informed consent impossible.
7. FEV 1/FVC < 50% of predicted, DLCO < 50% of predicted.
8. Resting LVEF < 50%.
9. Bilirubin > 2.0 mg/dl, transferase (AST) > 2x upper limit of normal, unless the abnormalities are secondary to Crohn's disease.
10. Serum creatinine > 2.0 mg/dl.
11. Platelet count less than 100,000/ul, ANC less than 1500/ul.
12. Patients presenting with intestinal perforation or toxic megacolon, or a suppurative problem that will require urgent surgery. In addition, the patient may not have any active infection. The presence of intestinal stomas does not exclude the patient from study.
13. Pre-study peripheral blood counts must include a platelet count greater than 100,000/ul and an absolute neutrophil count greater than 1500/ul.
14. Creatinine clearance more than 20% below lower limit of normal for age and sex.
15. Short gut syndrome.

Donor eligibility

Inclusion criteria

1. Donor must be an HLA 6 out of 6 matched sibling

Exclusion criteria of HLA matched sibling donor

1. Physiologic age > 50 years old or <18 years old
2. HIV positive
3. Active ischemic heart disease or heart failure
4. Acute or chronic active hepatitis
5. Uncontrolled diabetes mellitus or any other illness that in the opinion of the investigators would jeopardize the ability of the donor to tolerate stem cell collection
6. Prior history of malignancy except localized basal cell or squamous skin cancer. Other malignancies for which the patient is judged to be cured by local surgical therapy, such as (but not limited to) head and neck cancer, or stage I or II breast cancer will be considered on an individual basis.
7. Positive pregnancy test
8. Psychiatric illness or mental deficiency making compliance with treatment or informed consent impossible
9. Major hematological abnormalities such as platelet count less than 100,000/ul, ANC less than 1000/ul
10. Donor has history of Crohn's or ulcerative colitis

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2010-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Burt, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Allogeneic Stem Cell Therapy
Started | 9
Completed | 8
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Allogeneic Stem Cell Therapy
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.11 (7.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Survival
Description: The number of participants who survived treatment
Time Frame: Up to five years
Population: The number of participants who survived treatment
Measure: Number; unit: participants
Arm/Group | Allogeneic Stem Cell Therapy
Number analyzed (Participants) | 9
participants | 8

ADVERSE EVENTS:
Time Frame: Up to 5 years
Arm/Group | Allogeneic Stem Cell Therapy
All-Cause Mortality (participants affected / at risk) | 1/9
Serious Adverse Events (participants affected / at risk) | 1/9
Other Adverse Events (participants affected / at risk) | 7/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Allogeneic Stem Cell Therapy (N=9)
Adenovirus infection (Infections and infestations) | 1 (1) — One mortality due to adenovirus colitis, hepatitis, and fulminate liver failure.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Allogeneic Stem Cell Therapy (N=9)
Clostridium difficile infection (C-Diff) (Infections and infestations) | 2 (2) — One participant developed C-Diff infection one month after the transplant . Another participant developed C-Diff infection while inpatient for transplant. Both were treated with Flagyl and infections resolved.
Sinusitis (Infections and infestations) | 1 (1) — One participant was diagnosed with sinusitis four months after the transplant, treated with oral antibiotics and resolved.
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) — In one patient, who had prior history of Tacrolimus associated AKI (Acute Kidney Injury), post transplant was complicated by AKI. Renal biopsy showed chronic tubule-intestinal disease, started on hemodialysis.
Anorexia (Gastrointestinal disorders) | 2 (2) — While in the hospital for transplant, two patients had disease related anorexia requiring parenteral nutrition
Strep throat (Infections and infestations) | 1 (1) — One patient had strep throat resolved with oral antibiotics
Cholecystectomy (Surgical and medical procedures) | 1 (1) — One patient two months post transplant developed cholecystitis requiring cholecystectomy
perianal abscess (Gastrointestinal disorders) | 1 (1) — One patient had disease related perianal abscess during transplant. resolved with antibiotics and incision and drainage
perforated colon (Gastrointestinal disorders) | 1 (1) — one patient 14 months post transplant underwent surgery to remove stricture-- during surgery colon perforated-- surgery showed no evidence of crohns
anorexia nervosa (Psychiatric disorders) | 1 (1) — one patient had anorexia nervosa before HSCT--continued after HSCT

LIMITATIONS AND CAVEATS:
Small numbers of subjects enrolled

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes